CLINICAL TRIAL: NCT05425654
Title: Rituximab, Methotrexate, Procarbazine, Vincristine, Lenalidomide (RL-MPV) Followed by BBC (BCNU, Busulfan, Cyclophosphamide) High-dose Chemotherapy With Auto-HCT and Maintenance Therapy With Nivolumab in Newly Diagnosed Primary CNS Lymphoma
Brief Title: RL-MPV Followed by BBC HCT Using Autologous Stem Cells and Maintenance Therapy With Nivolumab for Newly Diagnosed PCNSL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: "CNS-2021"
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Primary CNS Lymphoma
MeSH Terms: interventions — Rituximab; Methotrexate; Vincristine; Procarbazine; Lenalidomide; Busulfan; Carmustine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RL-MPV + BBC/auto-HCT+ nivolumab (Experimental): Rituximab, methotrexate (MTX), procarbazine, vincristine and lenalidomide (RL-MPV). The peripheral blood stem cell (PBSC) harvest procedure will be performed after 2nd cycle of RL-MPV. High dose chemotherapy Busulfan, Thiotepa, and Cyclophosphamide. 3 months after auto-HSCT, maintenance therapy with nivolumab 3 mg/kg is started for 6 months every 2 weeks
  Interventions: Drug: Rituximab, Methotrexate, Vincristine, Procarbazine, Lenalidomide

INTERVENTIONS:
Drug: Rituximab, Methotrexate, Vincristine, Procarbazine, Lenalidomide — The initial treatment will consist of cycles of 14 days. Each cycle will start with rituximab, which will be given by vein on day 1. On day 2 you will receive: Methotrexate will be given by vein over 2 to 3 hours and vincristine will be given as a single injection over a few minutes. Procarbazine and Lenalidomide are a pill that you will take at bedtime for 7 nights starting on day 2. Procarbazine and Lenalidomide are only given every other cycle. During each cycle, you will be in the hospital. After the second cycle of chemotherapy, PBPCs will be collected. You will be hospitalized again for high-dose chemotherapy and receive supportive medications to help avoid complications, including antibiotics and blood transfusions. Busulfan, carmustine and cyclophosphamide will be given to you for 5 days. After break of 1 day, we will return your PBPC (or bone marrow) to you through a vein. You will be in the hospital for at least 3 weeks.
  Other Names: Busulfan, Carmustine, and Cyclophosphamide

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the new treatment proposed in this study. Conducting a prospective study "CNS-2015" in patients with PDLBCL CNS made it possible to achieve 2-year EFS, DFS and OS of 83%, 83% and 88%, respectively. The presence of early relapses of the disease has now led to the need to find an alternative program for patients with PDLBCL CNS. In the new "CNS-2021" protocol, lenalidomide was included in the R-MPV program in order to intensify the induction stage. In the conditioning regimen, thiotepa was replaced by carmustine, due to its significant CNS bioavailability. In order to possibly prevent early relapses, an anti-PD-1 inhibitor (nivolumab) was used as maintenance therapy.

DETAILED DESCRIPTION:
Patients will receive 4 cycles of RL-MPV (rituximab, methotrexate (MTX), procarbazine, vincristine, and lenalidomide (RL-MPV) as induction. The conditioning regimen prior to autologous blood stem cell transplantation includes high doses busulfan, thiotepa, and cyclophosphamide. After 3 months after autologous blood stem cell transplantation, maintenance therapy with nivolumab 3 mg/kg every 2 weeks for 6 months will be started.Patients will be out of the study at the time of death. All patients believe in the possibility of survival within 3 months throughout their lives. Survival status can be obtained by phone call, storage visit, or medical records (eg doctor's note/lab results from a clinic or storage visit).

ELIGIBILITY:
Inclusion Criteria:

All patients must have non-Hodgkin's lymphoma involving the brain, as demonstrated by CT or MRI and histologic confirmation by one of the following: A positive CSF cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers.

A biopsy of the vitreous or uvea demonstrating non-Hodgkin's lymphoma. Brain biopsy.

Patients must be HIV-1 negative. Patient must have left ventricular ejection fraction ≥ 50%. Patients must have no evidence of systemic lymphoma. This must be demonstrated by a CT scan of the chest, abdomen and pelvis prior to registration.

Patients must have adequate bone marrow function (defined as peripheral leucocyte count >3000 cells/mm3 and platelet count > 100,000 cells/mm3), liver function (bilirubin < 2.0 mg/%), and adequate renal function (serum creatinine < 1.5 mg/dl or creatinine clearance > 50cc/min/1.73M2).

Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.

Patients must be between 18 and 70years-old. Patients must sign an informed consent.

Exclusion Criteria:

Prior cranial irradiation Other active primary malignancy. Pre-existing immunodeficiency such as renal transplant recipient. Prior treatment with chemotherapy for CNS lymphoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
frequency of adverse events | Time Frame: 1-year event-free survival and acute treatment-related toxicity.]
  to evaluate the frequency of adverse events (safety and efficacy) of the use of RL-MPV followed by high-dose chemotherapy using carmustine, cyclophosphamide and busulfan with stem cell rescue in patients with newly diagnosed PCSNL.

SECONDARY OUTCOMES:
response rates | Time Frame: after 56 days (after 4 cycles - each cycle is equal to 14 days)
  to evaluate response rates with the combination of lenalidomide and R-MPV as induction chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nathional Medical Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No